CLINICAL TRIAL: NCT06364891
Title: Assessing the Impact of a Segment-targeted Mobilization Model Supported by a Digital VMMC Platform on Uptake of VMMC Services in Zambia
Brief Title: Assessing the Impact of a Digital VMMC Platform
Acronym: VMMC NEXUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Principal Investigator, Carolyn Bolton, Principle Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VMMC NEXUS; INV-047777 (Other Grant/Funding Number: Bill & Melinda Gates Foundation)
Record Dates: First submitted 2024-03-25; First posted 2024-04-15 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Voluntary Medical Male Circumcision

STUDY DESIGN:
Intervention Model Description: Cluster randomised control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Other): Mobilisers in the intervention sites will be trained to use a digital mobile application to assist with segmenting clients and providing them with targeted messaging.
  Interventions: Other: VMMC NEXUS Digital application
- Control (Other): Mobilisers in the control arm have been sensitised to the segmentation process but only have access to paper based resources.
  Interventions: Other: VMMC NEXUS Digital application

INTERVENTIONS:
Other: VMMC NEXUS Digital application — A handheld digital application which supports segmentation of potential VMMC Clients

SUMMARY:
VMMC has been identified as a crucial intervention by UNAIDS to achieve the 2030 global target of a 90% reduction in new HIV infections compared with 2010 levels. CIDRZ, a key partner to the Ministry of Health, has worked with DesireLine to develop a mobile application that supports mobilisers to segment potential clients and provide them with targeted messaging based on their segmentation type. The hypothesis of our proposed study is that targeted interventions addressing the barriers for each of the seven segments, assisted by the Digital Mobilization Tool, will better meet the needs of potential clients and therefore improve uptake of VMMC services, specifically among the three most-resistant segments.

The objective of this study is to evaluate the effect of a segment-targeted mobilization intervention supported by the VMMC NEXUS Digital Mobilization Tool on the uptake of VMMC services at 30 intervention sites, compared with 30 control sites.

The research questions are:

1. What is the effect of segment-targeted mobilization interventions designed to address the specific psycho-behavioral barriers each of the seven segments face, supported by the VMMC NEXUS Digital Mobilization Tool, on the overall numbers of men receiving VMMC in each site?
2. What is the effect of the same on the numbers of men by segment receiving VMMC in each site?
3. What is the effect of the same on the numbers of men by age receiving VMMC in each site?

Secondary goals will be the following, to the extent possible:

* Assess the incremental cost of the intervention, including by MC
* Assess and document process learnings from the intervention
* Develop a workplan to enable national and regional scale-up of the mobilization model and NEXUS Digital Mobilization Tool if demonstrated as effective

DETAILED DESCRIPTION:
Study design

The study is a cluster randomised study. Programmatic data will be collected at 60 health-facility sites offering VMMC:

* 30 sites randomly selected as intervention sites
* 30 sites randomly selected as control sites Mobilizers associated with the intervention sites will mobilize men for VMMC using the segment targeted interventions for all seven segments, supported by the VMMC NEXUS Digital Mobilization Tool. At the control sites, mobilizers will use the current standard of care tools to engage men for VMMC; these tools are not digital and do not contain the targeted messaging for the three most-resistant segments. One study-supported mobilizer will be placed in each of the 60 sites to support mobilization of men for VMMC in the intervention and control sites as described above.

Mobilizer Training and Specialization The 60 mobilizers (one for each site, control or intervention) will be compensated with a monthly stipend and all will be trained on the basics of VMMC as an HIV prevention method and active listening approaches to educating clients about VMMC.

Mobilizers at the 30 intervention sites additionally will be trained on the VMMC segmentation and barriers men face to getting VMMC. Also they will be trained on use of the VMMC NEXUS Digital Mobilization Tool and on outreach approaches to the three most-resistant segments of men. Data entered by the mobilizers supporting the intervention sites as a part of their routine use of the VMMC NEXUS Digital Mobilization Tool to support their mobilization efforts will be monitored by the CIDRZ program team. Ongoing oversight and support will be provided to all mobilizers as part of routine management for both control and intervention sites.

Site Selection In order to control for potential differences between implementing partners, the study will use only those sites currently receiving technical assistance from CIDRZ. To select sites, the investigators reviewed data on the aggregate monthly number of MCs performed over a 24-month period (October 2020 - September 2022) at 893 health facilities that receive technical support from CIDRZ, in four provinces. Selection focused on the most active facilities by first selecting the sites that had performed at least 10 MCs in at least 1 month within the 24-month period. This yielded 777 sites. Next, those sites that had performed at least 10 MCs monthly in at least 18 months of the 24-month period were selected. There were 131 of these sites. To further refine the eligibility criteria, within each province sites were divided into rural and urban settings. Within each of these 8 categories (4 provinces X 2 types of setting) sites that reached at least the 25th percentile of average monthly volume of MCs were selected. This ensured a representative sample of active rural and active urban sites within each province, accounting for the fact that the average MC volume varies by province and setting. These sites were then randomly assigned to the intervention group or the control group to be balanced between groups controlling for the following: volume of Shang Ring procedures, volume of surgical procedures, volume of each of the 7 segments, province proportions and urban-rural proportions.

Methodology The study will record the number of men being engaged by the intervention mobilization efforts vs. the number receiving VMMC will be used to evaluate "conversion rates," both overall and by segment. The VMMC NEXUS Digital Tablet Mobilization Tool will facilitate data collection and tracking for this metric.

For men coming into facilities for VMMC, a standardised intake form, which includes a segmenting tool, will be used to record which segment a man belongs to and other demographic data, including age. The intake form will also collect information on which interventions men were exposed to before coming to the facility for VMMC. These data will be aggregated across facilities in localities where study mobilizers are using the Digital Mobilization Tool (intervention sites), and facilities where mobilisers are using the current standard of care tools (control sites).

The study team will extract aggregated weekly data, including VMMC volume data by segment and age. These data will be tracked for up to 6 months before the intervention is launched, and then for a period of 9-12 months after, to determine whether the intervention sites produce a higher volume of MCs than the control sites, and whether MC volumes among the three more-resistant segments are higher at the intervention sites than at the control sites.

Process Evaluation To assess the fidelity of the implementation of the interventions a process evaluation will be completed, including qualitative one-on-one interviews of key stakeholders in the pilot implementation including a selection of individuals from the following stakeholder groups: CIDRZ Mobilizers - control & intervention sites, Other catchment area mobilizers - control & intervention sites, Clients - control and intervention sites, Data officers, CIDRZ implementation team, CIDRZ NEXUS platform team, Providers, Intake counselors, Site In-charges, MoH District & Province leaders, Sub-district coordinators, MoH national VMMC program leadership, Zambia VMMC TWG members.

The following areas of the implementation process will be covered in the interviews as appropriate for each stakeholder group: Mobilization tools, Mobilizer training and learning, Mobilization tool content and continuous improvement of content, Data collection, local area coordination and national coordination.

Costing Cost data for social marketing and demand mobilization interventions will be shared by the study team and compared to the same for control sites. Example fixed and variable costs for service delivery, e.g., provider salaries, will be used to estimate the effects of increased volumes on per overall per MC costs based on the interventions implemented.

Because there may be a difference in the number of interactions required between a mobilizer and a client prior to the client agreeing to proceed with MC, or the time required (number of minutes) per interaction, we will also utilize the following additional methods:

1. Mobilizer time tracking logbooks: all mobilizers will be asked to keep a logbook of their time for a four-week period. This is to be filled out each day and includes information about the clients mobilized, their segmentation and the time spent per client.
2. Mobilizer observations and interviews: researchers will observe a sample of mobilizers to better understand how they spend their time. We propose a sample of 3-4 mobilizers (sites) per province across all four study provinces, for a total number of 12-16 mobilizers (sites). Researchers will silently observe the mobilizers while they interact with clients for one day (from 8:00am-12:30pm) per site. While observing, researchers will complete a duplicate mobilizer logbook (see #1 above) for comparison, adding any relevant notes. The aim of the observation is to better understand how mobilizers interact with clients and to verify correct completion of the logbooks.

We will use the time tracking data combined with other study data to estimate the average number of interactions per client at intervention and control sites and the time per interaction. We will also compare this data with the number of clients who choose to proceed with MC.

Relevant information on site-by-site VMMC service delivery capacities and campaign activities will be collected on a weekly basis to control for these variables in subsequent analyses. The following information will be collected by site: # of Dorsal Slit Surgery provider-days in the 7-day week, # of Shang Ringy provider-days in the 7-day week, # of active CIDRZ mobilizer-days, # of active Non-CIDRZ mobilizer-days, # of MC incentives paid to non-CIDRZ mobilizers, # prisoner MCs, Stock out Shang Ring commodities, Shang Ring-related stockout details, Stock outs of other MC commodities, Dorsal Slit MC-related stockout details, Campaign week, Campaign activities, IEC materials posted or distributed in the catchment area, Notes and other comments.

ELIGIBILITY:
Inclusion Criteria:

living in the catchment area 18 or older

Exclusion Criteria:

nil

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150383 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Total number of VMMC's conducted in intervention vs control | at 12 months
  The study will compare the difference in total number of VMMC's conducted in the intervention versus the control arm
Total number of VMMC's by segment | at 12 months
  The total number of VMMC's conducted in both the intervention and control arm will be compared by segment (ie the specific group type the men have been assigned to).
Total number of VMMC's by age | at 12 months
  The total number of VMMC's conducted in both the intervention and control arm will be compared and stratified by age group.

SECONDARY OUTCOMES:
Costing | 12 months
  The study will assess the incremental cost of the intervention, including by MC
Process evaluation | 12 months
  The study will assess the fidelity of the intervention (ie how well the inertvention was implemented) and document all process learnings (ie opportunities and obstacles, changes that were required, unanticipated challenges etc) from the intervention
Develop a workplan and handbook to allow for the intervention to be scaled up elsewhere. | 3 months post study completion
  The study team will develop a template workplan and comprehensive scale up document to enable national and regional scale-up of the mobilization model and NEXUS Digital Mobilization Tool if demonstrated as effective

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health facilities, Lusaka, Lusaka Province, Zambia